CLINICAL TRIAL: NCT04389151
Title: Triplezumab Combined With CAPEOX Regimen Was Used in a Phase II Clinical Study of Neoadjuvant Therapy for Locally Advanced Colon Cancer With MSI-H /dMMR
Brief Title: Triplezumab Combined With CAPEOX Regimen in Neoadjuvant Therapy for Locally Advanced Colon Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JS001-ISS-CO24
Record Dates: First submitted 2020-04-28; First posted 2020-05-15 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-04

CONDITIONS: Locally Advanced Colon Cancer
MeSH Terms: interventions — toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The experimental group (Other)
  Interventions: Drug: Toripalimab

INTERVENTIONS:
Drug: Toripalimab — Toripalimab union CAPEOX scheme： Toripalimab 240mg, ivgtt, Q3w Oxaliplatin 130mg/m2,ivgtt, Q3w capecitabine 1000mg/m2, p.o Q3w

SUMMARY:
According to the 2019NCCN guidelines, immunocheckpoint inhibitors are recommended for first-line treatment of metastatic colon cancer patients with high microsatellite instability (msi-h) or mismatched gene deletion (dMMR) who are not suitable for intensive treatment, and for all patients with second-line or above msi-h /dMMR treatment.This study is a single-center, single-arm phase II study of the use of triplezumab (JS001) combined with CAPEOX regimen in the neoadjuvant therapy of msi-h /dMMR for locally advanced colon cancer. The subjects received neoadjuvant therapy with triplezumab (JS001) combined with CAPEOX regimen, with one treatment cycle every 3 weeks and two cycles of surgery followed by pathological evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Sign written informed consent.
2. Age ≥18 years.
3. ECOG physical condition score ≤1.
4. Pathological diagnosis of msi-h /dMMR colon cancer.
5. The TNM stage of colon cancer was ct3/4nxm0 or ctxn1/2m0.
6. Never received anti-tumor treatment including but not limited to radiotherapy, chemotherapy and surgery.
7. The patient must have adequate organ function and meet the following laboratory test values during the screening period within 7 days before enrolling:

   * Absolute neutrophil cell count (ANC) ≥1.5x109/L, platelet ≥100x109/L, hemoglobin ≥90g/L.(in (Patients with no blood transfusion or growth factor support should be given for 7 days prior to blood collection.)
   * Serum creatinine ≤1.5× upper normal range (ULN) or estimated creatinine clearance ≥50mL/min.
   * Total bilirubin ≤1.5×ULN;If there is Gilbert syndrome or if the indirect bilirubin concentration indicates an extrahepatic source of bile The rise of erythrosin is ≤3×ULN.
   * Glutamate aminotransferase and glutamate aminotransferase (AST and ALT)≤3×ULN.
   * Aptt ≤1.5×ULN, and INR or PT≤1.5×ULN.
8. Fertile women must be willing to participate in the final CAPEOX programme during the study period and in conjunction with the triplezumab (JS001) Contraceptive measures were taken at least 120 days after administration, and urine or serum pregnancy tests were negative for 7 days prior to enrollment.
9. Unsterilized male subjects must be willing to participate during the study and at the end of the triplezumab (JS001) combined CAPEOX regimen Use contraception for at least 120 days after the first dose.
10. Good compliance, agreed to cooperate with the survival follow-up.

Exclusion Criteria:

1. Signs of distant metastasis.
2. The presence of complete obstruction, massive bleeding, or perforation associated with a colon tumor.
3. Previous use of immunocheckpoint inhibitors targeting ctla-4, pd-1 or pd-l1.
4. Have radiotherapy plan before or after operation.
5. A history of research on drug ingredients and severe allergic reactions to any monoclonal antibody.
6. Severe infection in the active stage or poorly controlled clinically.
7. Symptomatic congestive heart failure (New York heart association grade ii-iv) or symptomatic, poorly controlled arrhythmia often; Any arterial thromboembolic events that occurred or occurred within 6 months prior to inclusion included myocardial infarction, unstable angina cerebrovascular accident or transient ischemic attack; Deep vein thrombosis, pulmonary embolism, or any other serious condition occurred 3 months prior to enrollment, History of thromboembolism (implantable venous infusion port or catheter-induced thrombosis, or superficial venous thrombosis is not seen severe thromboembolism).
8. Subjects with any active, known or suspected autoimmune disease.History of autoimmune disease, including but not limited myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis related to antiphospholipid syndrome, wegener's granulomatosis, sjogren's syndrome, guillain-barre complex signs, multiple sclerosis, vasculitis, or glomerulonephritis.
9. Patients with autoimmune hypothyroidism who receive stable dose hormone replacement therapy are eligible to participate in this study investigate.
10. Patients with vitiligo or who have had complete remission of childhood asthma may be included without any intervention in adulthood.
11. Asthma patients requiring intermittent use of bronchodilators, inhaled steroids, or topical injections were not excluded from the study outside.
12. Use of corticosteroids (>10mg/ day prednisone or equivalent) or other within 14 days prior to initial administration subjects who received systemic therapy with immunosuppressive agents.In the absence of active autoimmune disease, inhalation or topical administration of corticosteroids and adrenal hormone replacement at dose ≤10mg/ day of prednisone.
13. Subjects with highly suspected interstitial lung disease, or interstitial lung disease requiring steroid hormone therapy, or other severe cases were excluded diseases that seriously affect lung function.
14. Get a live vaccine 4 weeks before joining.
15. Patients with other active malignancies within 5 years prior to the first use of the study drug.Localized tumors that have been cured, such as skin basal cell carcinoma, skin squamous cell carcinoma, superficial bladder carcinoma, prostate carcinoma in situ, cervical carcinoma in situ, breast carcinoma in situ, etc into the group.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-03-04 (Actual); Primary Completion 2021-03-04 (Estimated); Study Completion 2021-03-04 (Estimated)

PRIMARY OUTCOMES:
effectiveness of neoadjuvant therapy | 6 weeks
  The main pathological response rate of neoadjuvant therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Yefeng, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: Undecided